CLINICAL TRIAL: NCT02682615
Title: Cardiac Output Monitoring System (esCCO™) in Comparison to Transcardiopulmonal Thermodilution Technique (PiCCO®) in Critically Ill Patients Within Interdisciplinary Surgical Intensive Care Units
Brief Title: Non-invasive Cardiac Output Monitoring (esCCO™) in Critically Ill Patients Within ICU
Status: Withdrawn | Type: Observational
Why Stopped: Due to problems regarding methodology.
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PD Dr., University Hospital Schleswig-Holstein
Other Study IDs: A138-15
Record Dates: First submitted 2016-01-12; First posted 2016-02-15 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Cardiac Output
Keywords: Cardiac Index; Noninvasive; esCCO; PiCCO; Thermodilution

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- requirement of norepinephrine: requirement of norepinephrine <0,1 µg/kgKG/min versus ≥0,1 µg/kgKG/min

SUMMARY:
Evaluation of a non-invasive technique to measure cardiac output (esCCO™) with the "clinical goldstandard" of the transcardiopulmonal thermodilution technique (PiCCO®). Effect of different potential interference factors to the accuracy of measurement (changing concentration of norepinephrine, generally severity of the basic disease - APACHE II score).

DETAILED DESCRIPTION:
The measurements have to estimate the agreement of esCCO™ and PiCCO® related to the cardiac output (cardiac index). It should consult a comparison of methods between a complete non-invasive cardiac output monitoring method (esCCO™) and the transcardiopulmonal thermodilution technique (PiCCO®). The accuracy shall carve out as well as the power of agreement of both measurement methods.

It takes two simultaneous measurements at a time of critically ill patients at interdisciplinary surgical intensive care units. Furthermore the force of the major variables (1. requirement of norepinephrine and 2. APACHE II-score) to the estimators shall be realized.

esCCO™ vs. (PiCCO®)

This research shall include 100 patients which have to undergo a complex intensive care treatment within predefined therapy intentions.

During a daily screening within the interdisciplinary surgical intensive care units of the Universitätsklinikum Schleswig-Holstein, Campus Kiel it will be opted for the inclusion of the patients.

Points of time x [x ε M and M = {1, 2, 3, 4}] - two test series (measurement 1 and 2).

According to the ability of the patient to the research the predefined point of time number 1 will be supposed (point of time number 1: inclusion criterium). The predefined point of time number 2 will be supposed if the therapy concept is planned or changed. The point of time number 3 is defined as the re-evaluation in the course of changed therapy conceptions. If the medical practitioner team decides to renounce the PiCCO-system, the predefined point of time number 4 has arrived.

The requirement of norepinephrine will be registered in every measurement (1 and 2). The APACHE II-score will be surveyed each point of time x (see above).

The remaining treatment of the patients will be performed in the conventional way by the medical practitioner team within the interdisciplinary surgical intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* The extended haemodynamic monitoring procedure PiCCO® has already been established due to the clinical decision making of the medical practitioner team

Exclusion Criteria:

* atrial fibrillation
* cardiac arrhythmias
* cardiac pacemaker
* intraaortic counterpulsation
* pericardial tamponade
* age < 18 years
* missing or incorrect patient consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is the estimation of the agreement between esCCO™ and the transcardiopulmonal thermodilution technique (PiCCO®) using Bland-Altman-treatment. The 95%-confidence interval of the limits of agreement was selected for the design of the number of cases. At a number of cases by 100 you will get the width of 0,68 s (s: standard deviation of the differences of the measurement techniques). This is reasonable for the question (Bland and Altman 1986, you have to compare the recommendation of Bland: https://www.users.york.ac.uk/~mb55/meas/sizemeth.htm).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between esCCOTM and the transcardiopulmonal thermodilution technique (PiCCO®) | through study completion, an average of 1 year
  Comparison of cardiac output, utilizing cardiac index (CI), between (esCCO™) and the "clinical goldstandard" of the transcardiopulmonal thermodilution technique (PiCCO®)

SECONDARY OUTCOMES:
Effect of different potential interference factors to the accuracy of measurement (changing concentration of norepinephrine, generally severity of the basic disease) | through study completion, an average of 1 year
  Comparison of cardiac output, utilizing cardiac index (CI), between (esCCO™) and the "clinical goldstandard" of the transcardiopulmonal thermodilution technique (PiCCO®)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, PD Dr. med, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- GERMANY - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No